CLINICAL TRIAL: NCT01989065
Title: Healthy Lifestyles Program for You (HLP4U): Augmenting Childhood Obesity Treatment Through Provider-to-parent Text Messaging.
Brief Title: Healthy Lifestyles Program for You (HLP4U): Augmenting Childhood Obesity Treatment.
Acronym: HLP4U
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00050555; Pro00050555_RDS
Record Dates: First submitted 2013-11-14; First posted 2013-11-20 (Estimated); Last update posted 2015-12-03 (Estimated); Status verified 2015-12

CONDITIONS: Pediatric Obesity
Keywords: Child obesity; childhood obesity; obesity treatment; text messaging; Lifestyle
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lifestyle counseling (Active Comparator): The Duke Healthy Lifestyles program is a comprehensive childhood obesity treatment program. Standard of care is active engagement and Lifestyle Counseling of families by nutritionist, physician, mental health provider, and physical therapist. Monthly visits for 1 year are recommended.
  Interventions: Behavioral: Lifestyle counseling
- Lifestyle counseling PLUS text messaging (Experimental): Patients in this arm will receive full standard of care as described for the Active Comparison group. In addition, parents will be texted daily with a motivational message that provides information and support for healthy behaviors.
  Interventions: Behavioral: Lifestyle counseling; Behavioral: Text Messaging

INTERVENTIONS:
Behavioral: Lifestyle counseling — see arm description
Behavioral: Text Messaging — See Arm Description
  Arms: Lifestyle counseling PLUS text messaging

SUMMARY:
Outpatient childhood obesity treatment has limited efficacy. This study aims to improve the health habits of parents of obese 5-12 year old children enrolled in the Duke Healthy Lifestyles Program by delivering educational and supportive text messages to the parent's mobile device.

DETAILED DESCRIPTION:
Protocol Title Healthy Lifestyles Program for You (HLP4U): Augmenting childhood obesity treatment through provider-to-parent text messaging.

Significance One in three children in the US are overweight or obese, a condition known to increase the risk of adult obesity and chronic disease. Behavioral treatment of pediatric and adolescent obesity is strongly recommended, and in research settings treatment has shown efficacy in reduction of child body mass index (BMI) and improved long-term health outcomes. However, clinical treatment models must operate within the constraints of the outpatient practice, and are limited in their ability to deliver the same intensity of intervention or outreach. Not surprisingly, clinic-based treatment of child obesity is less effective than in research settings.

"Motivational Interviewing" (MI) has emerged as a promising clinical method for improving health outcomes in childhood obesity treatment. "Motivation" is defined as an individual's expressed intention to change, and is divided into three measurable elements: importance, confidence, and readiness. The theoretical framework of MI focuses on the interpersonal aspects of behavioral change between patient and provider. MI emphasizes provider empathy, support for patient autonomy, exploring ambivalence and reinforcing change talk. Several studies have demonstrated that childhood obesity treatments that use MI effectively are more likely to achieve improved child outcomes than those who do not. These outcomes include decreased BMI,6 increased physical activity, and improvements in parental confidence.

The Healthy Lifestyles (HL) program is an AAP Stage 2-4 childhood obesity program3 located in Durham, NC. Children with BMI above the 95th percentile are referred to HL by their primary provider. The Healthy Lifestyles clinical protocol has been described elsewhere. In short, children aged 22 years and under with BMI ≥ 95th percentile are referred by their primary physician to the multidisciplinary HL clinic for treatment of obesity and related co-morbidities. The intervention involves monthly visits for one year to meet with medical, dietary, exercise and behavior specialists all certified in Motivational Interviewing. Despite the comprehensive model, and despite consistent delivery of behavior change counseling using motivational interviewing, the Healthy Lifestyles model does not lead to significant decreases in body mass index. Less than 25% of patients who initially enroll complete treatment. These outcomes are similar to other comprehensive child obesity programs nationally. There is a clear need for effective treatment options.

A rapidly evolving field of study is investigating the use of healthcare provider-to-text messages to augment patient behavior change. Text messaging is attractive, in part, because text penetrance to mixed ethnic, racial, and socioeconomic populations is high, and 80-81% of sent messages are read with a mean response time of 6 minutes. Text messages as simple reminders can lead to improvements in patient compliance with medications and immunizations. Text messages targeting behaviors can decrease TV viewing time among young children when texts are delivered to the parent. Text messages can also improve self-efficacy when they offer encouragement, recognize the difficulty of change, and congratulate the patient on change. To date, no studies have investigated the use of provider-to-parent text messages utilizing MI theory to increase the effectiveness of childhood obesity treatment.

Design A randomized, controlled, non-blinded clinical trial design will be utilized. The study team will identify qualifying parents as they arrive for their child's first scheduled clinic appointment to the Duke Healthy Lifestyles Program. The team has previously obtained IRB approval to approach Healthy Lifestyles families who qualify for research studies (Healthy Lifestyles Notification of Research, PRO00031251).

Study interventions A trained research assistant will collect all measures as described below, either through chart review or direct questioning of the parent. A registered nurse will collect the food recall measure (USDA) and perform the 3-minute step test; both are in accordance with current clinical protocol. Subjects will be randomized to the intervention or control group using a random number generator (Excel, 2010). Subjects randomized to the control group will receive usual care, which includes a lifestyle counseling visit, educational materials, and goal-setting by a physician and dietician, with follow up in 1 month. Subjects randomized to the intervention group will receive usual care as above PLUS daily text messages on their designated mobile device for four weeks. The content of the messages will provide information to parents on general health behaviors and offer supportive guidance. Text messages will be delivered through the use of an application (GoogleVoice) that is accessible to the investigator on a mobile or web-based system. The text message will be delivered directly to the parent's message inbox, and does not require the parent to download any software or applications. Patients may opt-out at any time by replying STOP to a text message. Rules for texting and opt-out instructions will be provided in writing. Subjects will be permitted to respond to the PI text. Subjects will be informed that the PI is not able to answer any medical, appointment, or treatment questions, and if asked, will reply with the office phone number for appropriate triage. An appointment reminder for the follow up visit will be texted to both intervention and control groups 2 days prior to the scheduled visit. Subjects will repeat a subset of measures at the time of presentation for care at the HL clinic at the follow up visit, or if they do not present for care, will be contacted by phone to complete the follow up measures.

ELIGIBILITY:
Inclusion Criteria:

* Adult aged 18 or older and is the child's primary caregiver ("parent")
* Child aged 5-12 years
* Child with age- and gender-specific BMI ≥ 95th percentile
* Parent has mobile phone with texting plan

Exclusion Criteria:

* Inability to read and write in English
* Parent with severe medical or mental health condition limiting ability to attend appointments
* Plan to move out of state in next 3 months

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 101 (Actual)
Dates: Start 2014-09; Primary Completion 2015-08 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Food and Activity Frequency Survey Score | 3 month post-enrollment
  Validated lifestyle behavior survey, addresses common behaviors such as beverages, fast food, television time. 20 questions on 4-point Likert.

SECONDARY OUTCOMES:
General Self-Efficacy Survey Score | 3 month post-enrollment
  Validated survey measures parental general self-efficacy. 10 questions on a 5-point Likert.

OTHER OUTCOMES:
Change in child's Body Mass Index | Baseline and 3-month
  Weight divided by the height squared. Gives indication of whether healthy lifestyle changes lead to short-term weight reduction.

CONTACTS AND LOCATIONS:
Overall Officials: Sarah C Armstrong, MD, Principal Investigator — Duke Health
Locations (1):
- Duke Children's Health Center, Durham, North Carolina, United States